CLINICAL TRIAL: NCT03940404
Title: Anlotinib Hydrochloride Therapy in Patients With Advanced Lung Cancer: A Real World Study.
Brief Title: Anlotinib Therapy in Patients With Advanced Lung Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Cttq (Industry)
Responsible Party: Sponsor
Other Study IDs: ALOT-LC1
Record Dates: First submitted 2019-04-27; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experiment: The patients whose treatment strategy containing anlotinib.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib will give orally, once daily on days 1-14 of a 21-day cycle. Dose reduction is allowed.
  Other Names: Other intervention depends on the patient's disease

SUMMARY:
Purpose of the study: To observe the efficacy and safety of Anlotinib Hydrochloric Therapy in Patients with advanced Lung cancer in real world.

Subjects of the study: advanced Lung cancer.

Methods of the study:

This is a real world, prospective, Non-Interventional, Follow-up registration study.

Patients will get Anlotinib according to their condition and willingness. Anlotinib will give orally, once daily on days 1-14 of a 21-day cycle. After the procedure, regular follow up after every cycle.

End point:

Primary end point: progression-free survival (PFS). Secondary end points: overall survival (OS), disease control rate (DCR), overall response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age, man or woman, who had to provide written informed consent prior to enrollment.
2. Patients who had to have histologically and/or cytologically confirmed NSCLC that failed at least 2 kinds of systemic chemotherapy (third line or beyond), or who will obtain benefit from antiangiogenic therapy after investigator's assessment.
3. Eastern Cooperative Oncology Group performance status of 0-2.

Exclusion Criteria:

1. Contraindication of anlotinib.
2. Pregnant or lactating women.
3. Other patients who can't enroll after investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced lung caner
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  progression-free survival

SECONDARY OUTCOMES:
OS | 1 year
  overall survival
ORR | 1 year
  overall response rate
DCR | 1 year
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- First People's Hospital of Hangzhou, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided